CLINICAL TRIAL: NCT06136429
Title: A Prospective, Multicenter, Single-arm Target-value Clinical Trial To Evaluate the Transcatheter Aortic Valve System Safety and Efficacy for the Treatment of Patients With Severe Aortic Stenosis
Brief Title: A Prospective, Multicenter, Single-arm Study to Evaluate a Transcatheter Aortic Valve System Safety and Efficacy for the Treatment of Patients With Severe Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pan Xiangbin (Other)
Responsible Party: Sponsor-Investigator, Pan Xiangbin, dean, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silara202301
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: The transcatheter aortic valve system consists of 7 parts, namely the valve, the delivery system, the catheter sheath, the exchange system, the recovery system, the development exchange solution, and the curing agent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR Treatment Group (Experimental)
  Interventions: Procedure: Transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: Transcatheter aortic valve replacement — Device: Transcatheter Heart Valve System (Silara SR)

SUMMARY:
Trial Title: Prospective, multicenter, single-arm target value clinical trial to evaluate the safety and efficacy of a transcatheter aortic valve system in the treatment of patients with severe aortic stenosis Test device: Transcatheter aortic valve system. Pilot Phase: Clinical Validation of Class III Medical Devices. Study design: prospective, multicenter, single-group target value. Sample size: 120 cases. Intended Use: The Transcatheter Aortic Valve System is indicated for patients with a diagnosis of severe aortic stenosis by the Comprehensive Heart Team.

Objective: This clinical trial is a prospective, multicenter, single-arm study to evaluate the safety and efficacy of the transcatheter aortic valve system in the treatment of patients with severe aortic stenosis.

Primary endpoint: 12-month postoperative all-cause mortality All-cause deaths include cardiac death and non-cardiac death. Secondary Endpoints: 1. Device success rate 2. Procedural success rate 3. Delivery system performance 4. Retrieval system performance (e.g. using a recycling system) 5. Exchange system performance 6. Valvular function at Immediately postoperative, 7 days/at discharge, 30 days, 6 months, 12 months, 2-5 years follow-up: valve stenosis, regurgitation, valve function (e.g., opening area, pressure gradient), paravalvular leakage 7. Improvement in quality of life at 30 days, 6 months, 12 months postoperatively 8. Improvement in cardiac function at 7 days/at discharge, 30 days, 6 months, 12 months, 2-5 years postoperatively

Experimental design:

This trial is a prospective, multicenter, single-group clinical study with a target value to evaluate the Transcatheter Aortic Valve system Safety and efficacy in the treatment of patients with severe aortic stenosis with 12 months of All-cause mortality after transcatheter aortic valve implantation.

The mortality rate was the primary study endpoint, and after statistical assumptions and sample size calculations, 120 patients were planned to be enrolled.

Patients were clinically followed immediately after valve implantation, 7 days postoperatively/at discharge, 30 days, 6 months, 12 months, and 2-5 years postoperatively.

In this trial, all relevant clinical data were collected, sorted out and statistically analyzed by an independent data management and statistics center and a clinical monitoring institution. All enrolled subjects underwent outpatient follow-up at 30 days, 6 months, and 12 months after surgery, and performed relevant imaging examinations (ultrasound, etc.) and laboratory tests and safety evaluations, and continuous follow-up and cardiac ultrasound examinations were performed annually at 2-5 years to observe the occurrence of adverse events to evaluate the long-term safety of the transcatheter aortic valve system.

The safety and efficacy of the transcatheter aortic valve system were evaluated with the subject's 12-month postoperative all-cause mortality as the primary endpoint, and the immediate postoperative device success rate, procedural success, retrieval system performance, valve function, cardiac function improvement, quality of life improvement, all-cause mortality in different follow-up periods, major adverse cardiovascular and cerebrovascular events, myocardial infarction, stroke, hemorrhage, acute kidney injury, permanent pacemaker implantation, serious vascular complications, and other TAVR-related complications were taken as the secondary endpoints to assist in evaluating the safety and efficacy of the test product, and to provide a basis for the final official listing and domestic marketing.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 70 years;
2. Patients with symptomatic severe aortic stenosis (mean pressure gradient across the aortic valve ≥ 40 mmHg (1 mmHg = 0.133 kPa) on echocardiography, or trans-aortic valve blood flow velocity ≥ 4.0 m/s, or aortic orifice area ≤ 1.0 cm2, or effective aortic orifice area index ≤0.6 cm2/m2)
3. NYHA Grading ≥ Level II;
4. Life expectancy of more than 1 year after implantation of the prosthetic valve;
5. Assessed by not less than two cardiothoracic surgeons, documented as a contraindication to surgery, or documented as unsuitable for conventional surgery;
6. Patients who can understand the purpose of the trial, voluntarily participate in and sign the informed consent form, and are willing to undergo relevant examinations and clinical follow-up.

Exclusion Criteria:

1. The imaging data shows that it is anatomically unsuitable for transcatheter aortic valve implantation;
2. Acute myocardial infarction (defined as Q-wave myocardial infarction, or non-Q-wave myocardial infarction with CK-MB≥ twice normal and/or elevated Tn (WHO definition)) occurring within 1 month before valve implantation);
3. Received any therapeutic traumatic cardiac surgery (other than coronary revascularization) within 1 month before valve implantation;
4. Implanted prosthetic heart valves at any location, or combined with other valves with severe stenosis or severe regurgitation;
5. Hemorrhagic constitution or coagulation dysfunction (platelet PLT<50×10^9/L);
6. Haemodynamic instability requiring continuous mechanical cardiac assistance;
7. Severe left ventricular dysfunction, left ventricular ejection fraction LVEF <20%;
8. Echocardiography shows intracardiac thrombosis or vegetation, etc.;
9. Renal insufficiency decompensation (endogenous creatinine clearance rate<20ml/min);
10. Active peptic ulcer or upper gastrointestinal bleeding within 3 months;
11. Cerebrovascular events (CVAs) within 3 months before valve implantation, excluding transient ischemic attack;
12. Allergy or contraindication to antiplatelet drugs, anticoagulant drugs, or contrast agents, resulting in the inability to perform preoperative or appropriate intraoperative medication, allergies, or contraindications to polymer materials;
13. Patients with active infective endocarditis or other active infections;
14. Concurrent participation in other drug or device studies.
15. In the opinion of the investigator, it is not suitable for enrollment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of All-cause Mortality [ Time Frame: 12 months ] Percentage of subjects who died from all causes in this population. | [ Time Frame: 12 months ]

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided